CLINICAL TRIAL: NCT02497287
Title: An Open-label, Long-term, Safety and Efficacy Study of Intranasal Esketamine in Treatment-resistant Depression
Brief Title: A Long-term, Safety and Efficacy Study of Intranasal Esketamine in Treatment-resistant Depression
Acronym: SUSTAIN-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CR107148; ESKETINTRD3004 (Other: Janssen Research & Development, LLC); 2014-004587-38 (EudraCT Number)
Record Dates: First submitted 2015-05-18; First posted 2015-07-14 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Treatment-resistant Depression
Keywords: Treatment-resistant Depression; Esketamine; Oral Antidepressant
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant | interventions — Esketamine; Duloxetine Hydrochloride; Antidepressive Agents; Escitalopram; Sertraline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Intranasal Esketamine plus oral antidepressant (Experimental): Open-Label Induction Phase: Participants will self-administer esketamine intranasally twice per week for 4 weeks as a flexible dose regimen (56 mg or 84 mg). Participants greater than or equal to (>=) 65 will start at a dose of 28 mg on Day 1. Direct-entry participants will initiate a new, open-label oral antidepressant (duloxetine, escitalopram, sertraline, or venlafaxine extended release [XR]) on Day 1; transferred-entry participants will continue the same oral antidepressant from ESKETINTRD3005. Optimization/Maintenance Phase: Participants will self-administer esketamine (56mg or 84mg for those < 65 years; 28 mg, 56 mg or 84 mg for those >= 65 years) intranasally once per week for 4 weeks; transferred entry responder subjects from ESKETINTRD3005 will start at a dose of 28 mg in the first week. All participants will continue their same oral antidepressant during this phase.
  Interventions: Drug: Esketamine (Intranasal Spray); Drug: Duloxetine (Oral Antidepressant); Drug: Escitalopram (Oral Antidepressant); Drug: Sertraline (Oral Antidepressant); Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant)

INTERVENTIONS:
Drug: Esketamine (Intranasal Spray) — Open-Label Induction Phase: Participants will self-administer esketamine intranasally twice per week for 4 weeks as a flexible dose regimen (56 mg or 84 mg for those < 65 years; 28 mg, 56 mg or 84 mg for those >= 65 years). Participants >= 65 years old will start at a dose of 28 mg on Day 1. Optimization/Maintenance Phase: Participants will self-administer esketamine intranasally (56 mg or 84 mg for those < 65 years; 28 mg, 56 mg or 84 mg for those >= 65 years) once weekly then individualized to either once weekly or once every other week based on the severity of depressive symptoms. Transferred-entry responder participants from ESKETINTRD3005 >= 65 years old will start at a dose of 28 mg in Week 5.
Drug: Duloxetine (Oral Antidepressant) — Duloxetine could be selected as the oral antidepressant medication by the investigator based on review of Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire (MGH-ATRQ) and relevant prior antidepressant medication information. The minimum therapeutic dose is 60 milligram per day (mg/day).
Drug: Escitalopram (Oral Antidepressant) — Escitalopram could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. The minimum therapeutic dose is 10 mg/day. Participants >= 65 years of age will be titrated up to 20 mg/day, but can lower the dose to 10 mg/day for tolerability.
Drug: Sertraline (Oral Antidepressant) — Sertraline could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Sertraline will be titrated up to a dose of 150 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 50 mg/day.
Drug: Venlafaxine Extended Release (XR) (Oral Antidepressant) — Venlafaxine Extended Release could be selected as the oral antidepressant medication by the investigator based on review of MGH-ATRQ and relevant prior antidepressant medication information. Venlafaxine Extended Release will be titrated for participants < 65 years of age up to a dose of 225 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 150 mg/day. For participants >= 65, it can be titrated up to a dose of 150 mg/day, but if not tolerated the dose can be reduced to the minimum therapeutic dose of 75 mg/day.

SUMMARY:
The purpose of this open-label, multicenter study is to assess the long term safety and efficacy of intranasal esketamine plus an oral antidepressant in participants with treatment-resistant depression (TRD).

DETAILED DESCRIPTION:
This is an open-label (the researchers and participants know the treatment the participant is receiving), multicenter (more than 1 study site), long-term safety and efficacy study of intranasal esketamine plus an oral antidepressant in participants with treatment-resistant depression (TRD). Participants will enter the study either directly (direct-entry participants) or after completing the Double-Blind Induction Phase of ESKETINTRD3005 (transferred-entry participants). The study consists of 4 phases: Screening Phase (4 weeks), Open-Label Induction Phase (4 weeks), Open-Label Optimization/Maintenance phase (48 weeks), and Follow up Phase (4 weeks). Transferred entry non-responders in the ESKETINTRD3005 may enter study at the Open-Label Induction Phase and responders in the ESKETINTRD3005 may enter Optimization/Maintenance phase. In the Open-Label Induction Phase, participants will self-administer flexibly-dosed intranasal esketamine (participants who are less than (<) 65 years old self-administer 56 mg or 84 mg dose, participants who are greater than or equal to (>=) 65 years old self-administer 28 mg, 56 mg or 84 mg dose) twice weekly for 4 weeks. The starting dose for all participants >= 65 years old will be 28 mg. In addition, each direct-entry participants will be assigned to receive 1 of 4 selected oral antidepressant medications (escitalopram or sertraline or duloxetine or venlafaxine extended release [XR]), initiated on Day 1 of the open-label induction phase and continued through the duration of the study. Transferred-entry participants will continue their same antidepressant from ESKETINTRD3005 through the duration of this study. Participants who are responders at the end of the Open-Label Induction phase and transferred-entry responder participants (from study ESKETINTRD3005) will enter the Optimization/Maintenance Phase where intranasal esketamine treatment sessions will be reduced from that in the induction phase (twice weekly) to weekly for the first 4 weeks of this phase, and then individualized to either once weekly or once every other week based on the severity of depressive symptoms. Participants' safety and depressive symptoms will be assessed and monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

A). For Direct-Entry Participants

* At the time of signing the informed consent form (ICF), participant must be a man or woman ≥18 (or older if the minimum legal age of consent in the country in which the study is taking place is greater than [>]18)
* At the start of the screening phase, participant must meet the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) (if single-episode MDD, the duration must be greater than or equal to [>=] 2 years) or recurrent MDD, without psychotic features, based upon clinical assessment and confirmed by the Mini-International Neuropsychiatric Interview (MINI)
* At screening, participant must have a MADRS total score of >=22
* At the start of the screening phase, participants must have had nonresponse to >=2 oral antidepressant treatments in the current episode of depression, as assessed using the the MGHATRQ and confirmed by documented records (example medical/pharmacy/prescription records or a letter from treating a physician, etc,) B). For Transferred-entry Participants
* All participants who completed the double-blind induction phase of ESKETINTRD3005 study, regardless of their response status, will be eligible to participate in this study, if they meet the study specific eligibility criteria

Exclusion Criteria:

A). For Direct-Entry Participants

* Participant's depressive symptoms have previously not responded to: Esketamine or ketamine in the current major depressive episode per clinical judgment or All of the 4 oral antidepressant treatment options available in the respective country for the open-label induction phase (that is, duloxetine, escitalopram, sertraline, and venlafaxine XR) in the current major depressive episode (based on Massachusetts General Hospital - Antidepressant Treatment Response Questionnaire [ MGH-ATRQ])
* Participant has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychotic features, bipolar or related disorders (confirmed by the MINI), obsessive compulsive disorder (current only), intellectual disability (DSM-5 diagnostic codes 317, 318.0, 318.1, 318.2, 315.8, and 319), autism spectrum disorder, borderline personality disorder, antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* Participant has homicidal ideation/intent, per the investigator's clinical judgment, or has suicidal ideation with some intent to act within 6 months prior to the start of the screening phase, per the investigator's clinical judgment or based on the Columbia Suicide Severity Rating Scale (C-SSRS)
* Participants with history of moderate or severe substance or alcohol use disorder according to DSM-5 criteria
* Participants who has a Mini Mental State Examination (MMSE) <25; Has neurodegenerative disorder (example, Alzheimer's disease, vascular dementia, Parkinson's disease), or evidence of mild cognitive impairment (MCI) B). Transferred-Entry Participants
* Participant has taken any prohibited therapies that would not permit dosing on Day 1

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2015-09-30 (Actual); Primary Completion 2017-10-28 (Actual); Study Completion 2017-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (109):
- United States (16):
  - New Haven, Connecticut
  - Miami, Florida
  - Marietta, Georgia
  - Iowa City, Iowa
  - Wichita, Kansas
  - Baltimore, Maryland
  - Watertown, Massachusetts
  - Cedarhurst, New York
  - New York, New York
  - Staten Island, New York
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - Wichita Falls, Texas
  - Richland, Washington
- Argentina (6):
  - Banfield
  - Buenos Aires
  - Córdoba
  - La Plata
  - Mendoza
  - Rosario
- Australia (4):
  - Adelaide
  - Caulfield
  - Frankston
  - Melbourne
- Austria (2):
  - Innsbruck
  - Vienna
- Belgium (2):
  - Bruges
  - Hasselt
- Brazil (7):
  - Belo Horizonte
  - Fortaleza
  - Recife
  - Rio de Janeiro
  - Santo André
  - São José do Rio Preto
  - São Paulo
- Bulgaria (9):
  - Burgas
  - Kardzhali
  - Kazanlak
  - Pazardzhik
  - Pleven
  - Plovdiv
  - Rousse
  - Sofia
  - Varna
- Finland (2):
  - Helsinki
  - Kuopio
- France (4):
  - Paris
  - Poitiers
  - Toulon
  - Tours
- Germany (3):
  - Berlin
  - Bochum
  - Oranienburg-Sachsenhausen
- Lithuania (3):
  - Kaunas
  - Šilutė
  - Vilnius
- Malaysia (3):
  - Ipoh
  - Johor Bahru
  - Kuala Lumpur
- Mexico (5):
  - Acapulco
  - Durango
  - Mexico City
  - México
  - Monterrey
- Gdansk, Poland
- South Africa (3):
  - Cape Town
  - Garsfontein
  - Pretoria
- South Korea (3):
  - Gwangju
  - Gyeonggi-do
  - Seoul
- Spain (9):
  - Badajoz
  - Bilbao
  - Madrid
  - Ourense
  - Oviedo
  - Sant Boi de Llobregat
  - Torrevieja
  - Valencia
  - Zamora
- Sweden (7):
  - Gothenburg
  - Halmstad
  - Lund
  - Skövde
  - Solna
  - Stockholm
  - Umeå
- Taiwan (6):
  - Kaohsiung City
  - New Taipei City
  - Taichung
  - Tainan
  - Taipei
  - Taoyuan
- Turkey (Türkiye) (6):
  - Ankara
  - Bursa
  - Gaziantep
  - Istanbul
  - Kocaeli
  - Manisa
- United Kingdom (8):
  - Bristol
  - Chesterfield
  - Derby
  - London
  - Middlesbrough
  - Northampton
  - Oxford
  - Preston

REFERENCES:
- [Derived] Oliveira-Maia AJ, Rive B, Godinov Y, Mulhern-Haughey S. Estimating the benefit of esketamine nasal spray versus real-world treatment on patient-reported functional remission: results from the ICEBERG study. Front Psychiatry. 2024 Oct 7;15:1459633. doi: 10.3389/fpsyt.2024.1459633. eCollection 2024. PMID 39435126
- [Derived] Oliveira-Maia AJ, Morrens J, Rive B, Godinov Y, Cabrieto J, Perualila N, Barbreau S, Mulhern-Haughey S. ICEBERG study: an indirect adjusted comparison estimating the long-term benefit of esketamine nasal spray when compared with routine treatment of treatment resistant depression in general psychiatry. Front Psychiatry. 2023 Oct 31;14:1250980. doi: 10.3389/fpsyt.2023.1250980. eCollection 2023. PMID 38025433
- [Derived] Oliveira-Maia AJ, Rive B, Morrens J, Godinov Y, Cabrieto J, Perualila N, Mulhern-Haughey S. Indirect adjusted comparison of 6-month clinical outcomes between esketamine nasal spray and other real-world polypharmacy treatment strategies for treatment resistant depression: results from the ICEBERG study. Front Psychiatry. 2023 Oct 31;14:1250987. doi: 10.3389/fpsyt.2023.1250987. eCollection 2023. PMID 38025416
- [Derived] Williamson D, Turkoz I, Wajs E, Singh JB, Borentain S, Drevets WC. Adverse Events and Measurement of Dissociation After the First Dose of Esketamine in Patients With TRD. Int J Neuropsychopharmacol. 2023 Mar 22;26(3):198-206. doi: 10.1093/ijnp/pyac081. PMID 36525338
- [Derived] Williamson DJ, Gogate JP, Kern Sliwa JK, Manera LS, Preskorn SH, Winokur A, Starr HL, Daly EJ. Longitudinal Course of Adverse Events With Esketamine Nasal Spray: A Post Hoc Analysis of Pooled Data From Phase 3 Trials in Patients With Treatment-Resistant Depression. J Clin Psychiatry. 2022 Sep 19;83(6):21m14318. doi: 10.4088/JCP.21m14318. PMID 36149841
- [Derived] Ochs-Ross R, Wajs E, Daly EJ, Zhang Y, Lane R, Lim P, Drevets WC, Steffens DC, Sanacora G, Jamieson C, Hough D, Manji H, Singh JB. Comparison of Long-Term Efficacy and Safety of Esketamine Nasal Spray Plus Oral Antidepressant in Younger Versus Older Patients With Treatment-Resistant Depression: Post-Hoc Analysis of SUSTAIN-2, a Long-Term Open-Label Phase 3 Safety and Efficacy Study. Am J Geriatr Psychiatry. 2022 May;30(5):541-556. doi: 10.1016/j.jagp.2021.09.014. Epub 2021 Oct 6. PMID 34750057
- [Derived] Wajs E, Aluisio L, Holder R, Daly EJ, Lane R, Lim P, George JE, Morrison RL, Sanacora G, Young AH, Kasper S, Sulaiman AH, Li CT, Paik JW, Manji H, Hough D, Grunfeld J, Jeon HJ, Wilkinson ST, Drevets WC, Singh JB. Esketamine Nasal Spray Plus Oral Antidepressant in Patients With Treatment-Resistant Depression: Assessment of Long-Term Safety in a Phase 3, Open-Label Study (SUSTAIN-2). J Clin Psychiatry. 2020 Apr 28;81(3):19m12891. doi: 10.4088/JCP.19m12891. PMID 32316080
- [Derived] Nijs M, Wajs E, Aluisio L, Turkoz I, Daly E, Janik A, Borentain S, Singh JB, DiBernardo A, Wiegand F. Managing Esketamine Treatment Frequency Toward Successful Outcomes: Analysis of Phase 3 Data. Int J Neuropsychopharmacol. 2020 Jul 29;23(7):426-433. doi: 10.1093/ijnp/pyaa027. PMID 32270176
- See also: An Open-label, Long-term, Safety and Efficacy Study of Intranasal Esketamine in Treatment-resistant Depression — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217051&parentIdentifier=CR107148&attachmentIdentifier=784eff25-9637-4962-8853-2319a9034a25&fileName=ESKETINTRD3004_(CR107148)_Additional_results_data_CH.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In this study participants from study ESKETINTRD3005 (NCT02422186) were enrolled (transferred entry [TE]). ESKETINTRD3005 is referred as TRD3005 in the draft.
Pre-assignment Details: Total 802 participants were enrolled (direct-entry [DE]=691 + TE from study ESKETINTRD3005 =111). Among 111 TE participants, 88 participants (non-responders from ESKETINTRD3005) joined induction (IND) phase and 23 participants (responders from ESKETINTRD3005) did not join IND phase and directly entered in optimization/maintenance (OP/MA) phase.
Groups:
- Intranasal Esketamine + Oral Antidepressant: Participants enrolled directly or TRD3005 non-responders self-administered intranasal Esketamine (Esk) twice a week for 4 weeks as age dependent flexible dose according to titration regimen for 56 or 84 milligram (mg) (<65 years) and 28, 56 or 84 mg (>=65 years) in IND phase. Participants who met response criteria at end of IND phase, entered OP/MA phase and received intranasal esketamine weekly from week 5-8 of OP/MA phase. From Week 9-52, participants received Esk either weekly or every other week based on MADRS score. TE (TRD3005 responders) joined OP/MA phase and received intranasal Esk 28, 56 or 84 mg weekly until week 8. DE participants initiated new oral antidepressant (AD) (1 of: duloxetine/escitalopram/sertraline/venlafaxine extended release [XR]) on Day 1 of IND phase and continued during IND and OP/MA phase. TE participants continued same oral AD from TRD3005. No intranasal Esk was given in follow-up phase and same oral AD was continued at investigator's clinical judgement.
Period: Induction Phase (4 Weeks)
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Started | 779 (Included DE participants (691) and non-responders from TRD3005 (88).)
Completed | 580
Not Completed | 199
Not completed — Did Not Met Criteria for OP/MA Phase | 84
Not completed — Adverse Event | 52
Not completed — Withdrawal by Subject | 22
Not completed — Lack of Efficacy | 21
Not completed — Other | 13
Not completed — Lost to Follow-up | 5
Not completed — Protocol Violation | 1
Not completed — Non-Compliance with Study Drug | 1
Period: Optimization/Maintenance (48 Weeks)
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Started | 603 (Included who completed IND phase (580) + responders from TRD3005 (23).)
Completed | 150
Not Completed | 453
Not completed — Study Terminated by Sponsor | 331
Not completed — Withdrawal by Subject | 30
Not completed — Adverse Event | 25
Not completed — Lack of Efficacy | 25
Not completed — Other | 21
Not completed — Lost to Follow-up | 10
Not completed — Protocol Violation | 3
Not completed — Missed Assessment or Treatment Sessions | 3
Not completed — Pregnancy | 2
Not completed — Death | 2
Not completed — Non-Compliance with Study Drug | 1
Period: Follow-up Phase (4 Week)
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Started | 357 (Included non-responders (IND phase) or discontinued treatment phase or completed OP/MA phase.)
Completed | 326
Not Completed | 31
Not completed — PI Decision | 12
Not completed — Withdrawal by Subject | 10
Not completed — Lost to Follow-up | 5
Not completed — Adverse Event | 3
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 802
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.2 (13.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 502
  Male | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 149
  Not Hispanic or Latino | 640
  Unknown or Not Reported | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 81
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 686
  More than one race | 8
  Unknown or Not Reported | 12
Region of Enrollment [Count of Participants; unit: Participants]
  ARGENTINA | 106
  AUSTRALIA | 23
  AUSTRIA | 16
  BELGIUM | 5
  BRAZIL | 52
  BULGARIA | 94
  FINLAND | 2
  FRANCE | 4
  GERMANY | 13
  ITALY | 7
  MALAYSIA | 19
  MEXICO | 10
  POLAND | 6
  SOUTH AFRICA | 64
  SOUTH KOREA | 26
  SPAIN | 42
  SWEDEN | 90
  TAIWAN | 33
  TURKEY | 31
  UNITED KINGDOM | 12
  UNITED STATES | 147

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event is any untoward medical occurrence in a clinical study participants who administered a medicinal (investigational or non-investigational) product and does not necessarily have a causal relationship with the treatment. A TEAE defined as an event that was new in onset or increased in severity following treatment initiation.
Time Frame: Up to End of Follow up Phase (Week 56)
Population: All enrolled analysis set included all transferred-entry and direct-entry participants who were not screen failures and received at least one dose of intranasal study medication or 1 dose of oral antidepressant.
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 802
Percentage of participants | 90.1

2. Primary Outcome: Percentage of Participants With Cystitis, Urinary Tract Infections, Renal and Urinary Tract Symptoms, Renal and Urinary Disorders
Description: Percentage of participants with cystitis, urinary tract infections, renal and urinary tract symptoms, renal and urinary disorders were evaluated. Cystitis and urinary tract infections are selected MedDRA preferred terms, "renal and urinary tract symptoms" refers to any preferred term (PT) in the group of selected PTs; and "renal and urinary disorders" refers to a MedDRA System Organ Class (SOC).
Time Frame: Up to End of Follow up Phase (Week 56)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 802
Percentage of participants
  Cystitis | 0.6
  Urinary tract infections | 8.1
  Renal and urinary disorders | 10.5
  Renal and urinary tract symptoms | 17.0

3. Primary Outcome: Change From Baseline in Cognitive Test Battery: Detection Test (DET) Score
Description: This battery is a series of computerized cognition tests (detection, identification, one card learning, one back and groton maze learning) designed to measure reaction time, visual learning and memory, and executive function/sequencing. The DET is a measure of psychomotor function and uses a well-validated simple reaction time. In this outcome measure, speed of performance of participants (calculated as mean of the logarithmic base 10 transformed reaction times) for correct responses was reported. Total score ranges from 2 to 3.3 log 10 milliseconds (msec). Lower score indicates better performance. Higher change from baseline indicates better performance.
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of Optimization/Maintenance [OP/MA] Phase)
Population: All enrolled analysis set included all transferred-entry and direct-entry participants who were not screen failures and received at least one dose of intranasal study medication or 1 dose of oral antidepressant. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: log10 msec
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 561
log10 msec | -0.0028 (0.12744)

4. Primary Outcome: Change From Baseline in Cognitive Test Battery: Identification Test (IDN) Score
Description: This battery is a series of computerized cognition tests (detection, identification, one card learning, one back and groton maze learning) designed to measure reaction time, visual learning and memory, and executive function/sequencing. IDN test is a measure of visual attention (choice reaction time) and scored for speed of response (mean of the log10 transformed reaction times for correct responses). Total score ranges from 2 to 3.3 log 10 msec. Lower score indicates better performance. Higher change from baseline indicates better performance.
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA Phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10 msec
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 561
log10 msec | -0.0083 (0.09656)

5. Primary Outcome: Change From Baseline in Cognitive Test Battery: One Card Learning Test (OCL) Score
Description: This battery is a series of computerized cognition tests (detection, identification, one card learning, one back and groton maze learning) designed to measure reaction time, visual learning and memory, and executive function/sequencing. OCL test is a measure of visual episodic memory and visual recall test scored using arcsine transformation of the percentage of correct responses (CR). The range for OCL is 0 to 100 percent (%) accuracy; presented as an arcsin transformation, the range is 0 to 1.57. Higher score indicates better performance. Higher change from baseline indicates better performance.
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA Phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Arcsine ([sqrt] of proportion of [CR])
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 561
Arcsine ([sqrt] of proportion of [CR]) | 0.0502 (0.13149)

6. Primary Outcome: Change From Baseline in Cognitive Test Battery: One Back Test (ONB) Score
Description: The ONB is a measure of working memory and scored for speed of correct response (mean of the log10-transformed reaction times for correct responses). Total score ranges from 2 to 3.54 log10 msec. Lower score indicates better performance. Higher change from baseline indicates better performance.
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA Phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: log10 msec
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 563
log10 msec | 0.0177 (0.10026)

7. Primary Outcome: Change From Baseline in Cognitive Test Battery: Groton Maze Learning Test (GMLT) Score
Description: This battery is a series of computerized cognition tests (detection, identification, one card learning, one back and groton maze learning) designed to measure reaction time, visual learning and memory, and executive function/sequencing. GMLT measures executive function; maze/sequencing test, scored for total number of errors. Total score ranges from 0 to 999 number of errors. Lower score indicates better performance. Higher change from baseline indicates better performance.
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA Phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of Errors
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 506
Number of Errors | 6.9 (25.36)

8. Primary Outcome: Change From Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) Score: Total Recall
Description: Hopkins Verbal Learning Test (HVLT) measures performance in verbal memory, learning, and long-term recall in which a list of words is read up to three times. Approximately 20-25 minutes later, a delayed recall trial and a recognition trial are completed. The delayed recall requires free recall of any words remembered. The recognition trial is composed of 24 words, including the 12 target words and 12 false-positives. When scoring the HVLT, the three learning trials are combined to calculate a total recall score (0-36); the delayed recall trial creates the delayed recall score (0 -12); the retention (%) score (0-100%) is calculated by dividing the delayed recall trial by the higher of learning trial 2 or 3; and the recognition discrimination index is comprised by subtracting the total number of false positives from the total number of true positives. A higher score = higher cognition.
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA Phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number correct
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 569
Number correct | 2.8 (4.74)

9. Primary Outcome: Change From Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) Score: Delayed Recall
Description: HVLT measures performance in verbal memory, learning, and long-term recall in which a list of words is read up to three times. Approximately 20-25 minutes later, a delayed recall trial and a recognition trial are completed. The delayed recall requires free recall of any words remembered. The recognition trial is composed of 24 words, including the 12 target words and 12 false-positives. When scoring the HVLT, the three learning trials are combined to calculate a total recall score (0-36); the delayed recall trial creates the delayed recall score (0 -12); the retention (%) score (0-100%) is calculated by dividing the delayed recall trial by the higher of learning trial 2 or 3; and the recognition discrimination index is comprised by subtracting the total number of false positives from the total number of true positives. A higher score = higher cognition.
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA Phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number correct
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 569
Number correct | 0.8 (2.31)

10. Primary Outcome: Change From Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) Score: Number of Words Recalled
Description: as for outcome 9
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA Phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of words recalled
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 568
Number of words recalled | 0.3 (2.83)

11. Primary Outcome: Change From Baseline in Hopkins Verbal Learning Test-Revised (HVLT-R) Score: Recognition Discrimination Index
Description: as for outcome 9
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA phase)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Number of words
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 568
Number of words | 0.5 (3.16)

12. Secondary Outcome: Change From Baseline to Endpoint in Montgomery Asberg Depression Rating Scale (MADRS) Total Score During Induction (IND) Phase
Description: MADRS measures depression severity, detects changes due to AD treatment. It consists 10 items (evaluate apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, suicidal thoughts), scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score of 0 to 60. Higher scores indicate more severe condition. Negative change in score indicates improvement. Missing data was imputed using last observation carried forward (LOCF) method, last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 4 weeks of IND phase)
Population: The full (IND) analysis set included all participants who received at least 1 dose of intranasal study medication or 1 dose of oral AD in open-label IND phase (for direct-entry and transferred-entry non-responder participants). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 756
Units on a Scale | -16.4 (8.76)

13. Secondary Outcome: Change From Baseline to Endpoint in MADRS Total Score During Optimization/Maintenance (OP/MA) Phase
Description: MADRS measure depression severity, detects changes due to AD treatment. It evaluates 10 items: apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, suicidal thoughts, each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score of 0 to 60. Higher scores represent a more severe condition. Negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Baseline (OP/MA) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA Phase)
Population: Full (OP/MA) analysis set: All participants who received at least 1 dose of intranasal study medication or 1 dose of oral AD in the OP/MA phase.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 603
Units on a Scale | 0.3 (8.12)

14. Secondary Outcome: Change From Baseline to Endpoint in Patient Health Questionnaire - 9 (PHQ-9) Total Score During IND Phase
Description: PHQ-9 is a 9-item, self-reporting scale assessing depressive symptoms. Each item was rated on a 4-point scale (0 = Not at all, 1 = Several Days, 2 = More than half the days, and 3 = Nearly every day), with a total score range of 0-27. A higher score indicates greater severity of depression. Severity of PHQ-9 categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), severe (20-27). The recall period is 2 weeks. Negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 4 weeks of IND phase)
Population: Full (IND) analysis set: All participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in the open-label IND phase (for direct-entry and transferred-entry non-responder participants). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Unit on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 746
Unit on a Scale | -8.9 (6.67)

15. Secondary Outcome: Change From Baseline to Endpoint in PHQ-9 Total Score During OP/MA Phase
Description: as for outcome 14
Time Frame: Baseline (OP/MA) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA phase)
Population: Full (OP/MA) analysis set: All participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in the OP/MA phase.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 603
Units on a Scale | -0.2 (5.65)

16. Secondary Outcome: Change From Baseline to Endpoint in Clinical Global Impression of Severity (CGI-S) Scale Score During IND Phase
Description: CGI-S measures severity of participant's illness that include knowledge of participant's history, psychosocial circumstances, symptoms, behavior, impact of symptoms on participant's ability to function. CGI-S evaluates severity of psychopathology on a scale range from 0 - 7, where 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. Negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as "Endpoint".
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 4 weeks of IND phase)
Population: Full (IND) analysis set: All participants who received at least 1 dose of intranasal study medication or 1 dose of oral AD in the open-label IND phase (for direct-entry and transferred-entry non-responder participants). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 763
Units on a Scale | -2.0 [-6 to 2]

17. Secondary Outcome: Change From Baseline to Endpoint in CGI-S Scale Score During OP/MA Phase
Description: The CGI-S measures the severity of the participant's illness that include knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S evaluates the severity of psychopathology on a scale of 0 to 7, where 0=not assessed; 1=normal (not at all ill); 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. Negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Baseline (OP/MA) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA phase)
Population: The full (OP/MA) analysis set included all participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in the OP/MA phase.
Measure: Median (Full Range); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 603
Units on a Scale | 0.0 [-3 to 4]

18. Secondary Outcome: Change From Baseline to Endpoint in Generalized Anxiety Disorder (GAD-7) Total Score During IND Phase
Description: GAD-7 is brief, validated 7-item self-reported assessment of overall anxiety. Participant's responded to each item using a 4 point scale with response categories: 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield total score ranges from 0 to 21, higher scores indicate more anxiety. Negative change in score indicates improvement. Severity of GAD-7 is categorized as: None (0-4), Mild (5-9), Moderate (10-14), Severe (15 -21). Missing data was imputed using LOCF method, last post baseline observation during the phase was carried forward as "Endpoint".
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 4 weeks of IND phase)
Population: The full (IND) analysis set included all participants who received at least 1 dose of intranasal study drug or 1 dose of oral AD in the open-label IND phase (for direct-entry and transferred-entry non-responder participants). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 724
Units on a Scale | -5.9 (5.85)

19. Secondary Outcome: Change From Baseline to Endpoint in GAD-7 Total Score During OP/MA Phase
Description: GAD-7 is brief and validated 7-item self-reported assessment of overall anxiety. Participants respond to each item using a 4 point scale with response categories: 0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day. Item responses are summed to yield a total score ranges from 0 to 21, higher scores indicate more anxiety. Negative change in score indicates improvement. Severity of the GAD-7 is categorized as follows: None (0-4), Mild (5-9), Moderate (10-14), Severe (15 -21). Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Baseline (OP/MA) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA phase)
Population: Full (OP/MA) analysis set: All participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in the OP/MA phase. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 574
Units on a Scale | 0.2 (4.23)

20. Secondary Outcome: Change From Baseline to Endpoint in European Quality of Life (EuroQol) 5-Dimension, 5-Level (EQ 5D-5L) During IND Phase: Sum Score
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ visual analogue scale (EQ VAS). EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a Health Status Index (HSI). HSI ranges from -0.148 to 0.949 and is anchored at 0 (health state value equal to dead) and 1 (full health). EQ VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 4 weeks of IND phase)
Population: The full (IND) analysis set included all participants who received at least 1 dose of intranasal study drug or 1 dose of oral AD in the open-label IND phase (direct-entry, transferred-entry non-responder participants). Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 745
Units on a Scale | -15.3 (16.26)

21. Secondary Outcome: Change From Baseline to Endpoint in EQ-5D-5L Score During IND Phase: EQ-VAS
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ VAS. EQ VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine).
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 4 weeks of IND phase)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 746
Units on a Scale | 17.0 (21.69)

22. Secondary Outcome: Change From Baseline to Endpoint in EQ-5D-5L Scale Score During IND Phase: Health Status Index
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a HSI. HSI ranges from -0.148 to 0.949 and is anchored at 0 (health state value equal to dead) and 1 (full health).
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 4 weeks of IND phase)
Population: as for outcome 20
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 745
Units on a Scale | 0.190 (0.2138)

23. Secondary Outcome: Change From Baseline to Endpoint in European Quality of Life (EuroQol) 5-Dimension, 5-Level (EQ 5D-5L) During OP/MA Phase: Sum Score
Description: EQ-5D-5L consists of EQ-5D-5L descriptive system and EQ VAS. EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each has 5 levels of perceived problems (1-no problem, 2-slight problems, 3-moderate problems, 4-severe problems, 5-extreme problems). Participant selects answer for each of 5 dimensions considering response that best matches his/her health "today". Responses were used to generate a Health Status Index (HSI). HSI ranges from -0.148 to 0.949 and is anchored at 0 (health state value equal to dead) and 1 (full health). EQ VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Sum score ranges from 0 to 100 where, sum score = (sum of the scores from the 5 dimensions minus 5) *5. Higher score indicates worst health state.
Time Frame: Baseline (OP/MA) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA phase)
Population: The full (OP/MA) analysis set included all participants who received at least 1 dose of intranasal study drug or 1 dose of oral AD in OP/MA phase.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 603
Units on a Scale | -0.7 (13.19)

24. Secondary Outcome: Change From Baseline to Endpoint in EQ-5D-5L Score During OP/MA Phase: EQ-VAS
Description: as for outcome 21
Time Frame: Baseline (OP/MA) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA phase)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 603
Units on a Scale | 1.6 (18.51)

25. Secondary Outcome: Change From Baseline to Endpoint in EQ-5D-5L Scale Score During OP/MA Phase: Health Status Index
Description: as for outcome 22
Time Frame: Baseline (OP/MA) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA phase)
Population: as for outcome 23
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 603
Units on a Scale | -0.009 (0.1411)

26. Secondary Outcome: Change From Baseline in Sheehan Disability Scale (SDS) Total Score During IND Phase
Description: SDS was a 5 item questionnaire used for assessment of functional impairment and associated disability. The first three items assess disruption of (1) work/school, (2) social life, (3) family life/home responsibilities using a 0 to 10 rating scale. Score for the first three items are summed to create a total score of 0 to 30, higher score indicates greater impairment and a negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Baseline (IND) up to the Endpoint (last post-baseline assessment value during 4 weeks of IND Phase)
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 626
Units on a Scale | -9.3 (7.86)

27. Secondary Outcome: Change From Baseline in Sheehan Disability Scale Total Score During OP/MA Phase
Description: SDS was a participant-reported outcome measure and was a 5 item questionnaire used for assessment of functional impairment and associated disability. The first three items assess disruption of (1) work/school, (2) social life, and (3) family life/home responsibilities using a 0 to 10 rating scale. The score for the first three items are summed to create a total score of 0 to 30 where a higher score indicates greater impairment and a negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Baseline (OP/MA) up to the Endpoint (last post-baseline assessment value during 52 weeks of OP/MA phase)
Population: The full (OP/MA) analysis set included all participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in the OP/MA phase. Here, 'N' (number of participants analyzed) signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 541
Units on a Scale | -1.6 (8.25)

28. Secondary Outcome: Percentage of Participants With Response as Assessed by MADRS Total Score During IND Phase
Description: Response is defined as greater than or equal to (>=) 50 % reduction from baseline in the MADRS total score. MADRS measures depression severity, detects changes due to AD treatment. It consists 10 items (evaluate apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, suicidal thoughts), scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score of 0 to 60. Higher scores indicate more severe condition. Negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Days 8, 15, 22 and Endpoint (last post-baseline assessment during 4 weeks of IND phase)
Population: The full (IND) analysis set included all participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in the open-label IND phase (for direct-entry and transferred-entry non-responder participants). Here, 'n' signifies those participants who were evaluable at specific time point for this endpoint.
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 779
Percentage of participants
  Day 8: number analyzed (Participants) | 739
  Day 8 | 11.6
  Day 15: number analyzed (Participants) | 751
  Day 15 | 25.0
  Day 22: number analyzed (Participants) | 753
  Day 22 | 42.8
  End point: number analyzed (Participants) | 756
  End point | 78.4

29. Secondary Outcome: Percentage of Participants With Response as Assessed by PHQ-9 Total Score During IND Phase
Description: Response is defined as >= 50 % reduction from baseline (IND phase) in PHQ-9 total score. PHQ-9 is a 9-item, self-reporting scale assessing depressive symptoms. Each item was rated on a 4-point scale (0 = Not at all, 1 = Several Days, 2 = More than half the days, and 3 = Nearly every day), with a total score range of 0-27. The scores are summed for a total score ranging from 0-27. A higher score indicates greater severity of depression. Severity of PHQ-9 categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), severe (20-27). The recall period is 2 weeks. Negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Day 15 and Endpoint (last post-baseline assessment value during 4 Week IND phase)
Population: The full (IND) analysis set included all participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in the open-label IND phase (for direct-entry and transferred-entry non-responder participants). Here, 'n' signifies those participants who were evaluable at specific time point for this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 779
Percentage of participants
  Day 15: number analyzed (Participants) | 724
  Day 15 | 37.2
  End point: number analyzed (Participants) | 744
  End point | 62.0

30. Secondary Outcome: Percentage of Participants With Remission as Assessed by MADRS Total Score During IND Phase
Description: Remission is defined as MADRS total score less than or equal to (<=) 12. MADRS measures depression severity, detects changes due to AD treatment. It consists 10 items (evaluate apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, suicidal thoughts), scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), summed for a total possible score of 0 to 60. Higher scores indicate more severe condition. Negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Days 8, 15, 22 and Endpoint (last post-baseline assessment value during 4 weeks of IND Phase)
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 779
Percentage of participants
  Day 8: number analyzed (Participants) | 739
  Day 8 | 7.3
  Day 15: number analyzed (Participants) | 751
  Day 15 | 15.6
  Day 22: number analyzed (Participants) | 753
  Day 22 | 27.2
  End point: number analyzed (Participants) | 756
  End point | 47.2

31. Secondary Outcome: Percentage of Participants With Remission as Assessed by PHQ-9 Total Score During IND Phase
Description: Remission is defined as PHQ-9 total score <= 4. PHQ-9 is a 9-item, self-reporting scale assessing depressive symptoms. Each item was rated on a 4-point scale (0 = Not at all, 1 = Several Days, 2 = More than half the days, and 3 = Nearly every day), with a total score range of 0-27. The scores are summed for a total score ranging from 0-27. A higher score indicates greater severity of depression. severity of PHQ-9 categorized as follows: none-minimal (0-4), mild (5-9), moderate (10-14), moderately severe (15-19), severe (20-27). The recall period is 2 weeks. Negative change in score indicates improvement. Missing data was imputed using LOCF method and the last post baseline observation during the phase was carried forward as the "Endpoint".
Time Frame: Day 15 and Endpoint (last post-baseline assessment value during 4 weeks of IND phase)
Population: as for outcome 29
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 779
Percentage of participants
  Day 15: number analyzed (Participants) | 726
  Day 15 | 12.7
  Endpoint: number analyzed (Participants) | 746
  Endpoint | 26.9

32. Secondary Outcome: Percentage of Participants With an Increase Score From Predose at Any Time in Clinician-Administered Dissociative States Scale (CADSS) Total Score During IND Phase
Description: The CADSS used to measure present-state dissociative symptoms, and to assess treatment-emergent dissociative symptoms. It comprises 23 subjective items divided into 3 components: depersonalization (with score range from 0 to 28), derealization (with score range from 0 to 52), and amnesia (with score range from 0 to 8). Participants responses are coded on a 5-point scale (0 = "Not at all", 1 = "Mild", 2 = "Moderate", 3 = 'Severe" and 4 = "Extreme"). The total score is sum of the 23 items and range from 0 to 92, where 0 (best) and 92 (worst). A higher score indicates a more severe condition.
Time Frame: Predose, up to 1.5 hours postdose (up to end of IND phase [Week 4])
Population: as for outcome 12
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 775
Percentage of participants | 92.0

33. Secondary Outcome: Percentage of Participants With an Increase Score From Predose at Any Time in CADSS Total Score During OP/MA Phase
Description: as for outcome 32
Time Frame: Predose, up to 1.5 hours postdose (up to end of OP/MA phase [Week 52])
Population: as for outcome 17
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 603
Percentage of participants | 86.1

34. Secondary Outcome: Percentage of Participants With Treatment-Emergent Acute Hypertension (Systolic and Diastolic) During IND and OP/MA Phases
Description: Percentage of participants with treatment-emergent acute hypertension (Systolic Blood Pressure >=180 millimeters of mercury [mm Hg] or Diastolic Blood Pressure >= 110 mm Hg) during IND and OP/MA Phases were evaluated.
Time Frame: Up to End of OP/MA phase (Week 52)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Intranasal Esketamine + Oral Antidepressant
Number analyzed (Participants) | 802
Percentage of participants
  Systolic BP >=180 | 2.2
  Diastolic BP >=110 | 2.4
  Acute hypertension | 4.1

ADVERSE EVENTS:
Time Frame: Up to follow up phase (Week 56)
Description: Population analyzed included all participants who received at least 1 dose of intranasal study medication or 1 dose of oral antidepressant in the respective phase (Induction, optimization or maintenance) and all participants who entered the follow-up phase.
Groups:
- IND: Intranasal Esketamine + Oral AD: Participants enrolled directly or TRD3005 non-responders self-administered intranasal Esk twice a week for 4 weeks as age dependent flexible dose according to titration regimen for 56 or 84 mg (age < 65 years) and 28, 56 or 84 mg (age >=65 years) in IND phase. DE participants initiated new oral AD (1 of: duloxetine/escitalopram/sertraline/venlafaxine XR) on Day 1 of IND phase. TE participants continued same oral AD from TRD3005.
- OP/MA: Intranasal Esketamine + Oral AD: Participants who met response criteria at end of IND phase, entered OP/MA phase and received intranasal Esk from Week 5-8 of OP/MA phase at same dose as in IND phase. From Week 9-52, participants received Esk either weekly or every other week depending on MADRS score. TE (TRD3005 responders) joined OP/MA phase and received intranasal Esk 28, 56 or 84 mg weekly until week 8. DE participants continued oral AD (1 of: duloxetine/escitalopram/sertraline/venlafaxine XR) same as in IND phase during OP/MA phase. TE participants continued same oral AD from TRD3005.
- FU: Intranasal Esketamine + Oral AD: Participants received no intranasal esketamine and continued same oral AD at the investigator's clinical judgement during 4-week follow-up (FU) phase.
Arm/Group | IND: Intranasal Esketamine + Oral AD | OP/MA: Intranasal Esketamine + Oral AD | FU: Intranasal Esketamine + Oral AD
All-Cause Mortality (participants affected / at risk) | 0/779 | 2/603 | 0/357
Serious Adverse Events (participants affected / at risk) | 17/779 | 38/603 | 8/357
Other Adverse Events (participants affected / at risk) | 587/779 | 454/603 | 24/357
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | IND: Intranasal Esketamine + Oral AD (N=779) | OP/MA: Intranasal Esketamine + Oral AD (N=603) | FU: Intranasal Esketamine + Oral AD (N=357)
Cardiac Failure Acute (Cardiac disorders) | 0 | 1 | 0
Anal Incontinence (Gastrointestinal disorders) | 0 | 1 | 0
Colitis Microscopic (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0
Large Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Oesophageal Ulcer (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0
Hepatitis Alcoholic (Hepatobiliary disorders) | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1 | 0
Dengue Fever (Infections and infestations) | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Hepatitis B (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 0 | 1 | 0
Pyelonephritis Acute (Infections and infestations) | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 0
Costochondral Separation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fibula Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Foot Fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0
Toxicity to Various Agents (Injury, poisoning and procedural complications) | 0 | 1 | 0
Transaminases Increased (Investigations) | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Neoplasm Malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 1 | 0
Psychomotor Hyperactivity (Nervous system disorders) | 1 | 0 | 0
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0
Alcohol Abuse (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Completed Suicide (Psychiatric disorders) | 0 | 1 | 0
Delirium (Psychiatric disorders) | 0 | 1 | 0
Delusion (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 5 | 3 | 5
Depression Suicidal (Psychiatric disorders) | 1 | 0 | 0
Intentional Self-Injury (Psychiatric disorders) | 0 | 1 | 0
Major Depression (Psychiatric disorders) | 1 | 0 | 0
Suicidal Ideation (Psychiatric disorders) | 2 | 4 | 0
Suicide Attempt (Psychiatric disorders) | 4 | 2 | 1
Stress Urinary Incontinence (Renal and urinary disorders) | 0 | 1 | 0
Tubulointerstitial Nephritis (Renal and urinary disorders) | 0 | 1 | 0
Vesical Fistula (Renal and urinary disorders) | 0 | 1 | 0
Menorrhagia (Reproductive system and breast disorders) | 0 | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | IND: Intranasal Esketamine + Oral AD (N=779) | OP/MA: Intranasal Esketamine + Oral AD (N=603) | FU: Intranasal Esketamine + Oral AD (N=357)
Vertigo (Ear and labyrinth disorders) | 68 | 43 | 1
Vision Blurred (Eye disorders) | 49 | 25 | 0
Diarrhoea (Gastrointestinal disorders) | 27 | 39 | 2
Hypoaesthesia Oral (Gastrointestinal disorders) | 63 | 28 | 0
Nausea (Gastrointestinal disorders) | 157 | 84 | 2
Vomiting (Gastrointestinal disorders) | 56 | 45 | 2
Fatigue (General disorders) | 40 | 28 | 1
Influenza (Infections and infestations) | 4 | 40 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 8 | 35 | 3
Urinary Tract Infection (Infections and infestations) | 26 | 48 | 7
Viral Upper Respiratory Tract Infection (Infections and infestations) | 19 | 70 | 1
Blood Pressure Increased (Investigations) | 53 | 46 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 14 | 33 | 1
Dizziness (Nervous system disorders) | 228 | 135 | 1
Dizziness Postural (Nervous system disorders) | 54 | 41 | 1
Dysgeusia (Nervous system disorders) | 77 | 54 | 0
Headache (Nervous system disorders) | 137 | 114 | 4
Hypoaesthesia (Nervous system disorders) | 79 | 40 | 0
Paraesthesia (Nervous system disorders) | 46 | 26 | 1
Sedation (Nervous system disorders) | 51 | 29 | 0
Somnolence (Nervous system disorders) | 94 | 85 | 0
Anxiety (Psychiatric disorders) | 49 | 26 | 1
Dissociation (Psychiatric disorders) | 182 | 113 | 1
Insomnia (Psychiatric disorders) | 40 | 34 | 1

LIMITATIONS AND CAVEATS:
Protocol defined study will be completed when at least 300 participants reach 26 weeks and 100 reach 52 weeks of treatment with esketamine. Discontinuation due to "Study terminated by sponsor" reflects reaching these prespecified completion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested in writing, such publication will be withheld for up to an additional 60 days.

DOCUMENTS (2):
  • Study Protocol (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/87/NCT02497287/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/87/NCT02497287/SAP_001.pdf